CLINICAL TRIAL: NCT00212966
Title: Shared Mental Health Care Linking General Hospital Acute Care Mental Health Services With Two Comprehensive Family Medicine Groups
Brief Title: Shared Mental Health Care Linking Mental Health Services With Family Medicine Groups
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: J. Robert Swenson, Ottawa Hospital Research Institute
Other Study IDs: 200334201H
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2010-08-23 (Estimated); Status verified 2010-08

CONDITIONS: Psychosocial Factors
Keywords: psychosocial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess how a multidisciplinary team of mental health professionals provides services to patients from two family medicine practices.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred by family physicians

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: family practice patients
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2004-07; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Swenson, MD, Principal Investigator — OHRI
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada